CLINICAL TRIAL: NCT04171544
Title: Streamline Occipito-Cervico-Thoracic System Post-Market Clinical Follow-up (OCT PMCF)
Brief Title: Streamline Occipito-Cervico-Thoracic System Post-Market Clinical Follow-up
Acronym: OCT PMCF
Status: Completed | Type: Observational
Sponsor: RTI Surgical (Industry)
Responsible Party: Sponsor
Other Study IDs: 1108-CL
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Spinal Stenosis Occipito-Atlanto-Axial; Spinal Disease; Spinal Stenosis Cervical; Spinal Stenosis Cervicothoracic Region; Spinal Instability
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Streamline Occipito-Cervico-Thoracic Spinal Fixation System — Spinal Fixation
  Other Names: Streamline OCT

SUMMARY:
This is a multi-center, post-market, retrospective study design to collect safety and performance data for patients implanted with the Streamline OCT System.

DETAILED DESCRIPTION:
This is a multi-center, post-market, retrospective study design to collect safety and performance data for patients implanted with the Streamline OCT System. The study will include a minimum of 58 patients at a minimum of 3 sites in the United States. The study will enroll at a minimum of 5 subjects implanted with the occipital plate.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have had an implant of the OCT System.

Exclusion Criteria:

* No exclusion criteria.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Subjects implanted with the OCT System.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Evaluate time to demonstration of fusion. | 12 months
  Evaluate time to demonstration of fusion.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Las Vegas Neurosurgical Institute, Las Vegas, Nevada
  - Spine Nevada, Reno, Nevada

IPD SHARING:
Plan to Share IPD: No